CLINICAL TRIAL: NCT00155220
Title: Treatment of Lymphedema- Application of the Kinesio Taping
Brief Title: Treatment of Lymphedema: Application of the Kinesio Taping
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9261701436
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-01-27 (Estimated); Status verified 2004-08

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Athletic Tape

INTERVENTIONS:
Device: Low Stretch Bandage and Kinesio Tape

SUMMARY:
There are 2 parts to this study.

First part:

* Reliability of water displacement, circumference, tonometer.
* Effect of taping: lifting effect measured with sonography
* Effect of taping: peripheral circulation measured with DRT4

Second part:

* Effects of different intervention models including decongestive lymphatic therapy (DLT) and modified DLT

DETAILED DESCRIPTION:
First part:

To investigate the reliability study of water displacement and circumference measurement and the change in thickness of subcutaneous space measured by sonography and blood flow measured by DRT4 in normal subjects after applying K-tape.

Second part:

The incidence of breast carcinoma is in the second place in women in Taiwan. Lymphedema is a common complication after treatment of breast carcinoma; it will lead not only to cosmetic problems but is also uncomfortable, and causes functional limitation for patients. The common management for lymphedema is decongestive lymphatic therapy (DLT) including skin care, manual lymph drainage, remedial exercises and compression therapies. At present, all possible compression therapies for lymphedema have limitations. Patients have poor compliance in using short-stretch bandage and compression garments due to the climate in Taiwan. Applying kinesio tape (K-tape) became a new treatment method in physical therapy; the inventor Dr. Kase claimed that the K-tape can improve circulation and remove congestion. Besides, it demonstrated good therapeutic effects in clinical application. However, there are few studies to show the clinical effects of K-tape. This restricts the further application of K-tape. Following the previous study, the purpose is to compare the effects among traditional DLT, modified DLT which replaces bandage with K-tape, and DLT combined K-tape in patients with lymphedema.

A randomized control study will be executed. Sixty patients with post-mastectomy lymphedema will be randomly grouped into taping, bandage and mixed groups. Each subject will go through 4 weeks of a control period, 4 weeks of an intervention period, and followed by 3 months of an observation period. The evaluation items include physical therapy assessment, the severity of swelling, such as arm circumference, volume of water displacement, related symptoms, the upper extremity function and quality of life. The evaluation will be executed 4 weeks before the interventions (start of control period), before the intervention (start of intervention period), after a 4 week intervention and 3 months after the intervention to compare the effects among 3 kinds of treatment. Subjects in each group will receive treatments including skin care, manual lymphatic drainage, pneumatic compression therapy and exercise during the intervention period; the taping group's patients will receive additional K-tape treatment; the mixed group's patients will receive K-tape combined bandage treatment. Each group will be treated 2 hours/time, 5 times/week; the entire course will take 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer lymphedema
2. Unilateral lymphedema
3. Lymphedema onset 3 months ago
4. Moderate to severe lymphedema
5. At least one measurement point greater than 2 cm
6. Good compliance

Exclusion Criteria:

1. Port-a-cath on affected side of chest with adhesion
2. Skin disease
3. Restriction of active range of motion
4. Affected upper extremity (UE)
5. Other diseases or medication might lead to swelling
6. Irremovable bracelet or ring

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-08; Study Completion 2006-03

PRIMARY OUTCOMES:
The severity of swelling, such as arm circumference, volume of water displacement
The evaluation will be executed 4 weeks before the interventions, before the intervention, after 4 week intervention and 3 months after intervention.

SECONDARY OUTCOMES:
Related symptoms, the upper extremity function and quality of life
The evaluation time the same as primary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Yih Tsauo, PhD, Study Chair — NTUH
Locations (1):
- School and Graduate Institute of Physical Therapy College of Medicine, National Taiwan University, Taipei, Taiwan